CLINICAL TRIAL: NCT06245590
Title: Evaluation of Low-dose Albumin and Midodrine Versus Midodrine Alone in Outcome of Recurrent Ascites in Patients With Decompensated Cirrhosis - An Open Label Multicentric Randomized Controlled Trial.
Brief Title: Evaluation of Low-dose Albumin and Midodrine Versus Midodrine Alone in Outcome of Recurrent Ascites in Patients With Decompensated Cirrhosis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-58
Record Dates: First submitted 2024-01-05; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-06

CONDITIONS: Decompensated Cirrhosis
MeSH Terms: interventions — Albumins; Midodrine; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Albumin + Midodrine (Experimental): Albumin + Midodrine (5mg thrice daily and will be increased every 3 days upto 15 mg thrice daily with target MAP (>75 mm and <90).
  Interventions: Drug: Albumin; Drug: Midodrine
- Midodrine +standard of care (Active Comparator): Midodrine alone titrated based on MAP.
  Interventions: Drug: Midodrine; Other: Standard of Care

INTERVENTIONS:
Drug: Albumin — 20 grams/ week Albumin + Midodrine (5mg thrice daily and will be increased every 3 days upto 15 mg thrice daily with target MAP (>75 mm and <90).
  Arms: Albumin + Midodrine
Drug: Midodrine — Midodrine
Other: Standard of Care — Standard of Care
  Arms: Midodrine +standard of care

SUMMARY:
The project is about evaluation of albumin and midodrine versus midodrine alone in outcome of recurrent ascites in patients with decompensated cirrhosis.

Cirrhosis occcurs in 50% of patients over 10 years. The mortality is approximately 40% at 1 year and 50% at 2 years (12.7 per 100,000 population). A lot of times the prognosis is poor and the main factors leading to it are - acute kidney injury, hepatorenal syndrome, hyponatremia, grade of ascites-recurrent ascites, sarcopenia, low mean arterial pressure.

Post review of the literature, it is realized that there are some gap areas -

* It is unknown whether combination of vasoconstrictor with albumin versus vasoconstrictor alone is superior for ascites resolution in patients with recurrent ascites.
* There are no studies till date on using combination of vasoconstrictor with albumin versus vasoconstrictor alone in patients with recurrent ascites.
* There are no studies on impact of combining vasoconstrictor and albumin in preventing the development of AKI and chronic kidney disease in these patients.

In an effort to bridge these gap areas, this project works on the following hypothesis - "Midodrine would have a synergistic effect with albumin in improving the systemic hemodynamics and circulatory dysfunction and will cause rapid control of ascites, reduce the incidence of large volume paracentesis (LVP), complications, reduce the incidence of chronic kidney disease (HRS-CKD) and improve outcome of patients with recurrent ascites in patients with decompensated cirrhosis as compared to midodrine alone"

Primary objective: To assess the effect of midodrine alone vs. a combination of midodrine and albumin on the survival free of TIPS and liver transplant at 6 months

Secondary objective:

The effect of midodrine alone vs. combination of midodrine and albumin on the cumulative frequency of therapeutic paracentesis at 6 and 12 months Proportion of patients achieving control of ascites at 6 and 12 months

DETAILED DESCRIPTION:
* Study population: Consecutive patients with decompensated cirrhosis with recurrent ascites seen as inpatients or outpatients in the Department of Hepatology at Institute of Liver and Biliary Sciences, who meet the inclusion criteria and provide informed consent
* Study design: Multicentre Open-label Randomised Controlled Trial
* Sample Size: Assuming that survival rate with albumin and midodrine is 80%, whereas with midodrine alone is 50% (i.e. 30% absolute difference is observed with alpha of 5% power, beta of 80%) we need to enroll 43 cases in each arm and taking 15% drop out rate we need to enrol 50 cases in each group.
* Intervention: Group A will be treated with 20 grams/ week Albumin + Midodrine (5mg thrice daily and will be increased every 3 days upto 15 mg thrice daily with target MAP (>75 mm and <90) and Group B midodrine alone titrated based on MAP. Albumin infusions will be provided with large volume paracentesis and if the patient develops AKI, SBP in the recommended dosage in accordance to the International Club of ascites. The protocol will be followed for 6 months

Adverse effects: Allergic reactions to albumin, worsening of dyspnea, volume-overload

Stopping Rule: adverse reaction to Albumin

* Cardiopulmonary compromise
* Allergic reaction

ELIGIBILITY:
Inclusion Criteria:

1. 18 -70yr and Cirrhosis with recurrent ascites.

Exclusion Criteria:

1. Recent Gastrointestinal bleeding within 7 days
2. Systemic arterial hypertension (>160/90mmhg)
3. Presence of hepatocellular carcinoma or portal vein thrombosis, Budd-chiari syndrome.
4. Pregnancy
5. No use of drugs affecting systemic hemodynamics (excepting beta blockers) 7 days prior to enrolment.
6. Patients with Cardiovascular disease (NYHA > II) or chronic obstructive pulmonary disease
7. Refusal to participate
8. Known or suspected hypersensitivity to albumin
9. Prior TIPS
10. Post liver or kidney transplantation
11. Patients enrolled in other clinical trials
12. Extrahepatic malignancy
13. Patients on cardiac glycosides like digoxin, phenylephrine, ephedrine, thyroid hormones, ergot derivatives, salt retaining steroids like fludrocortisone, MAO inhibitors, alpha blockers metformin and ranitidine (known to have interactions with midodrine)
14. Patients with intrinsic kidney disease, organ nephropathy and CKD stage 4 and
15. MELD > 25 and extremely moribund patient
16. Serum albumin less than 2 gm/dl or >3.5 gm/dl
17. Significant ongoing alcohol with abstinence less than 3 months
18. Significant findings on ECHO with cardiac dysfunction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-10 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Survival free of transplant and TIPS at 6 months. | 6 months

SECONDARY OUTCOMES:
The cumulative mean of the number of therapeutic paracentesis at 6 and 12 months would be compared between the two groups. | 6 & 12 months
Proportion of patients achieving resolution of ascites (complete grade 1-0 without diuretics and partial as garde 0-1 ascites on diuretics) | 6 & 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Asian Institute of Gastroenterology, Somājigūda, Hyderabad
  - Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi

IPD SHARING:
Plan to Share IPD: Undecided